CLINICAL TRIAL: NCT04785378
Title: The Effect of Use of Medical Masks on Exercise Capacity and Lower Extremity Endurance in Youth
Brief Title: The Effect of Use of Medical Masks on Exercise Capacity and Leg Endurance in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Meryem BEKTAŞ KARAKUŞ, Research Assistant, Acibadem University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09.2021.39
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Healthy Young People
Keywords: exercise capacity; medical mask; lower extremity endurance; youth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental)
  Interventions: Device: Medical mask; Other: Field tests

INTERVENTIONS:
Device: Medical mask — Participants will carry out field tests one day wearing a medical mask and the other day without a mask.
Other: Field tests — Participants will perform 6 MWT and ISWT tests to determine their exercise capacity, and a 30-second sit and stand test to determine lower extremity endurance.

SUMMARY:
The use of masks has become an important part of life in outbreak conditions. In order to prevent the spread of the outbreak, many people in society may have to wear masks for hours during the day. As a mask type, the medical mask is frequently preferred in society. There are limited studies on how the use of medical masks affects the person wearing the mask while performing various activities that require different energy needs during the day. Therefore, this study aims to investigate how the use of medical mask affects exercise capacity and leg endurance with simple field tests.

DETAILED DESCRIPTION:
Medical masks in use today are disposable and consist of three or four fine to very fine fibers. Medical masks are divided into three groups as type I, type II, and type IIR according to performance requirements. It is generally recommended for type I patients, type II, and type IIR healthcare professionals. The fact that many people in society use medical masks for hours in the current outbreak conditions and it is not known how long this situation will last suggests that the effects of the medical mask should be investigated further. This study was designed to investigate the effects use of a medical mask on exercise capacity and lower extremity endurance in young people. In the analysis using the G * Power 3.1.9.7 program, the sample size was calculated as 79 when the power ratio was at least 85% and the alpha error rate was 0.05. Participants included in the study will perform 3 field tests. Tests will be performed in the form of 30 seconds sit-to-stand test, incremental shuttle walk test (ISWT), and 6-minute walk test (6 MWT), respectively. Participants will come to the working place for 2 days to be evaluated. In this process, they will perform field tests one day with a medical mask and the other day without a mask. Whether the field tests to be performed on the first day will be with or without a medical mask will be decided through randomization. The tests to be made in the second visit will be carried out within 10 days with the time of the previous test, environmental conditions, and test sequence. The mask to be used in tests is a type I medical mask recommended for general public health in outbreak situations. The mask has three layers. During the study, the mask will be replaced with a new one at the end of each test. Also, mask-wearing comfort at rest, during daily living activities, and after ISWT will be evaluated with a 10-item scale. In the study, attention will be paid to precautions such as the researcher's use of a face shield and the protection of social distance in order to prevent the risk of contamination.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Not having any known acute/chronic diseases, especially respiratory, cardiac, and orthopedic pathologies
* HES code suitability (The HES code provides information about the covid-19 status of the person and is compulsorily questioned at the entrance to the institution where the study will be conducted.)

Exclusion Criteria:

* Presence of deformation in the face area that prevents the use of masks
* Individuals allergic to mask material

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
6 Minutes Walking Distance (6 DWD) | Until the second field tests are completed, up to 10 days
  6 MWD means the distance traveled in 6 MWT. Its unit is meters.
Distance traveled in ISWT | Until the second field tests are completed, up to 10 days
  It means the distance traveled in ISWT. Its unit is meters.
30 seconds sit to stand test result | Until the second field tests are completed, up to 10 days
  The result is the total number of stands within 30 seconds.

SECONDARY OUTCOMES:
Mask comfort level | Until the second field tests are completed, up to 10 days
  It is the evaluation of each of the 10 sensations that can occur with the use of a mask with visual analog scale (VAS).
Dyspnea VAS score | Until the second field tests are completed, up to 10 days
  It will be evaluated using VAS.
Dispnea modified borg scale (MBS) score | Until the second field tests are completed, up to 10 days
  It will be evaluated MBS.
Fatigue VAS score | Until the second field tests are completed, up to 10 days
  It will be evaluated using VAS.
Fatigue MBS score | Until the second field tests are completed, up to 10 days
  It will be evaluated using MBS.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Yıldız Özer, Assoc. prof., Study Director — Marmara University; Hızır Kurtel, Prof., Study Director — Marmara University; Meryem Bektaş Karakuş, Principal Investigator — Acıbadem Mehmet Ali Aydınlar University
Locations (1):
- Acıbadem Mehmet Ali Aydınlar University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Epstein D, Korytny A, Isenberg Y, Marcusohn E, Zukermann R, Bishop B, Minha S, Raz A, Miller A. Return to training in the COVID-19 era: The physiological effects of face masks during exercise. Scand J Med Sci Sports. 2021 Jan;31(1):70-75. doi: 10.1111/sms.13832. Epub 2020 Sep 30. PMID 32969531
- [Background] Fikenzer S, Uhe T, Lavall D, Rudolph U, Falz R, Busse M, Hepp P, Laufs U. Effects of surgical and FFP2/N95 face masks on cardiopulmonary exercise capacity. Clin Res Cardiol. 2020 Dec;109(12):1522-1530. doi: 10.1007/s00392-020-01704-y. Epub 2020 Jul 6. PMID 32632523
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Li Y, Tokura H, Guo YP, Wong AS, Wong T, Chung J, Newton E. Effects of wearing N95 and surgical facemasks on heart rate, thermal stress and subjective sensations. Int Arch Occup Environ Health. 2005 Jul;78(6):501-9. doi: 10.1007/s00420-004-0584-4. Epub 2005 May 26. PMID 15918037
- [Background] Person E, Lemercier C, Royer A, Reychler G. [Effect of a surgical mask on six minute walking distance]. Rev Mal Respir. 2018 Mar;35(3):264-268. doi: 10.1016/j.rmr.2017.01.010. Epub 2018 Feb 1. French. PMID 29395560
- [Background] Shaw K, Butcher S, Ko J, Zello GA, Chilibeck PD. Wearing of Cloth or Disposable Surgical Face Masks has no Effect on Vigorous Exercise Performance in Healthy Individuals. Int J Environ Res Public Health. 2020 Nov 3;17(21):8110. doi: 10.3390/ijerph17218110. PMID 33153145